CLINICAL TRIAL: NCT00310986
Title: Breathing Meditation With Methylphenidate for the Treatment of Attention Deficit Hyperactivity Disorder Children: A Randomized Controlled Trial
Brief Title: Breathing Meditation With Methylphenidate for the Treatment of Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE490230
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; meditation; breathing meditation; Anapanasathi; randomized controlled trial; nonpharmacologic treatment; complementary and alternative medicine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Behavioral: Breathing Meditation

SUMMARY:
In 2004, the Developmental Clinic of the Child Psychiatric Unit at Srinagarind Hospital, had 80 new pediatric cases of attention deficit hyperactivity disorder (ADHD) come for evaluation and intervention. The children were between 7-12 years of age. Most of them were treated with stimulant medication, (i.e. methylphenidate) to help reduce hyperactivity; however, both the parents and children needed special help to develop some techniques for behavioural management.

Meditation has been used as an attention training method for many thousands of years, and was mostly involved with religious or spiritual practices in various parts of the world, especially in the eastern countries. Breathing meditation is a popular method which can be applied to all people without instructions that are too complicated. If meditation therapy, by breathing meditation which is specified to treat attention deficit hyperactivity disorders, benefits this group of patients, it would be very useful, culturally appropriate, cost-effective and would reduce the drugs used which will save the child from drug side effects.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is the most common psychiatric disorder in children, with an estimated prevalence of 3-7% in school children (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision [DSM-IV-TR]). The major symptoms of this disorder are developmentally inconsistent and chronic levels of inattention, impulsiveness, and hyperactivity.

The numbers of patients visiting physicians for ADHD are increasing from year to year. Boys are diagnosed with ADHD three times more often than girls. Although the studies on adolescents are few, the data suggest that about half of the children diagnosed with ADHD will have persistent symptoms into adolescence and some symptoms persist into adulthood.

The symptoms of ADHD, if not adequately managed, will have many life long effects on the patients, families, friends, peers, teachers and colleagues. For the patients, the disorder will impact on patient's academic, social and emotional performance, and behavioural development, leading to poor academic achievement, low occupational status, increased risk of substance abuse and delinquency. More than 30% of children with ADHD repeat a year in school and up to 56% require remedial tutoring.

Drug therapy began in the 1930s; since the 1970s, stimulants such as dexamphetamine, and methylphenidate have increasingly been used as the treatment of choice, but remain controversial. Currently available psychological treatments for ADHD include behavioural training for teachers and parents, and parenting skills classes, behavioural therapy for children with ADHD. Psychosocial treatments are generally combined with medication because each treatment alone has only a partial effect on the core symptoms of the disorder.

Growing scientific evidence, clinical experience and community attitudes are encouraging a shift to more natural and holistic forms of therapy as alternatives or adjuncts to pharmacological approaches in a variety of conditions. Meditation has a wide range of applications, but it is especially useful in treating stress and related disorders to promote calmness and enhance the attentional ability. A psychological oriented definition stated that meditation is a set of attentional practices leading to an altered state or trait of consciousness characterized by expanded awareness, greater presence, and a more integrated sense of self.

Breathing Meditation could be classified as both concentrative meditation and mindfulness meditation. The concentrative ability is first developed at the beginning state and followed by mindful ability.

The studies which use meditation therapy for ADHD are still scarce. In Thailand, Hassasiri A, et al (1995) had developed meditation program for children with ADHD based on Neo-humanist concept which comprised of meditation and imagery . The program was tested in pre-post test design with purposive sampling and yielded the statistical significant different at p < 0.05 (unpublished data). There has never been research about the effectiveness of breathing meditation. We are interested in conducting a randomized controlled trial to study the effectiveness in patients with attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ADHD by a child psychiatrist using DSM-IV-TR criteria
* Any religious background
* Age between 7-12 years.
* Voluntariness and can adhere to the program

Exclusion Criteria:

* Autistic spectrum disorders
* Mental retardation

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-12 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Conners' Abbreviated Parent Questionnaire (continuous outcome) assessed by the parents at baseline, end of 4-week , at 8 weeks, and at 12 weeks

SECONDARY OUTCOMES:
Child Attention Problems (CAP) Rating Scale at the same time
Drugs used throughout 12 weeks program

CONTACTS AND LOCATIONS:
Overall Officials: Thawatchai Krisanaprakornkit, MD, Principal Investigator — Department of Psychiatry, Faculty of Medicine , Khon Kaen University
Locations (1):
- Department of Psychiatry, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Jensen PS, Kenny DT. The effects of yoga on the attention and behavior of boys with Attention-Deficit/ hyperactivity Disorder (ADHD). J Atten Disord. 2004 May;7(4):205-16. doi: 10.1177/108705470400700403. PMID 15487477
- [Result] Krisanaprakornkit T, Krisanaprakornkit W, Piyavhatkul N, Laopaiboon M. Meditation therapy for anxiety disorders. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004998. doi: 10.1002/14651858.CD004998.pub2. PMID 16437509
- [Result] Scahill L, Schwab-Stone M. Epidemiology of ADHD in school-age children. Child Adolesc Psychiatr Clin N Am. 2000 Jul;9(3):541-55, vii. PMID 10944656
- [Result] Barrows KA, Jacobs BP. Mind-body medicine. An introduction and review of the literature. Med Clin North Am. 2002 Jan;86(1):11-31. doi: 10.1016/s0025-7125(03)00069-5. PMID 11795084
- [Result] Mannuzza S, Klein RG, Bessler A, Malloy P, LaPadula M. Adult psychiatric status of hyperactive boys grown up. Am J Psychiatry. 1998 Apr;155(4):493-8. doi: 10.1176/ajp.155.4.493. PMID 9545994
- See also: The Khon Kaen University Ethics Committee for Human research — http://eckku.kku.ac.th/
- See also: Faculty of Medicine , KhonKaen University , Thailand — http://www.md.kku.ac.th/site_en/